CLINICAL TRIAL: NCT06711523
Title: A Phase III Clinical Study of the Efficacy and Safety of Polyethylene Glycolized Human Granulocyte Stimulating Factor Injection (PEG-G-CSF) in Preventing Neutropenia After Chemotherapy
Brief Title: Study Evaluating PEG-G-CSF Injectionin Preventing Neutropenia After Chemotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kexing Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KXZY-KB201702-301
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-11

CONDITIONS: Neutropenia, Chemotherapy-Induced Febrile; Breast Neoplasm Female
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.) (Experimental): A single subcutaneous injection of 6 mg PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.) was administered 24h+2h after the end of chemotherapy administration on day 1 of each chemotherapy cycle; Inject at least 1 cycle of chemotherapy with PEG-G-CSF injection, and up to 4 cycles of chemotherapy.
  Interventions: Drug: PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.)
- PEG-G-CSF injection (Neulasta®，Amgen Europe B.V.) (Active Comparator): Single subcutaneous injection of 6 mg PEG-G-CSF injection ( Neulasta®, Amgen Europe B.V.) 24h+2h after the end of chemotherapy administration on day 1 of each chemotherapy cycle in the abdomen (5 cm beyond the umbilicus); Inject at least 1 cycle of chemotherapy with PEG-G-CSF injection, and up to 4 cycles of chemotherapy.
  Interventions: Drug: PEG-G-CSF injection (Neulasta®，Amgen Europe B.V.)

INTERVENTIONS:
Drug: PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.) — This trial was conducted using the IWRS system where subjects were randomly assigned to the test group (PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.)) and control group (Neulasta®，Amgen Europe B.V.) in a 1:1 ratio.
  Arms: PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.)
Drug: PEG-G-CSF injection (Neulasta®，Amgen Europe B.V.) — This trial was conducted using the IWRS system where subjects were randomly assigned to the test group (PEG-G-CSF injection (Kexing Biopharmaceutical Co., Ltd.)) and control group (Neulasta®，Amgen Europe B.V.) in a 1:1 ratio.
  Arms: PEG-G-CSF injection (Neulasta®，Amgen Europe B.V.)

SUMMARY:
To evaluate the efficacy, safety, and immunogenicity of PEG-G-CSF Injection (Kexing Biopharmaceutical Co., Ltd.) for the prevention of neutropenia after chemotherapy, using the PEG-G-CSF Injection ( Neulasta®, Amgen Europe B.V.) as a positive control.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤75 years
2. Female breast cancer patients with a pathohistologically confirmed diagnosis requiring first-time adjuvant or neoadjuvant chemotherapy and for whom the following regimens are appropriate: ① EC regimen (epirubicin 90 mg/m2 iv day 1, cyclophosphamide 600 mg/m2 iv day 1) ② TC regimen (cyclophosphamide 600 mg/m2 iv day 1, docetaxel 75 mg/m2 iv day 1) ③ TCb regimen ( docetaxel 75 mg/m2 iv day 1, carboplatin AUC=5 iv day 1); Note: TCb regimens such as the combination of anti-HER2 targeting drugs H (trastuzumab) and P (pertuzumab) can also be included.
3. Physical condition ECOG score ≤ 1;
4. Weight ≥ 45kg;
5. Peripheral blood cell counts eligible for chemotherapy: white blood cell (WBC) count ≥ 3.5 x 109/L, neutrophil count (ANC) ≥ 1.5 x 109/L, hemoglobin (HB) ≥ 90 g/L, platelet (PLT) count ≥ 100 x 109/L, normal coagulation or abnormalities of no clinical significance, and no tendency to bleed;
6. Survival is expected to be 6 months or more;
7. The subject is willing to use an appropriate method of contraception for the duration of the trial;
8. Subjects agreed to follow the trial treatment protocol and visit schedule, enrolled voluntarily, and signed a written informed consent form.

Exclusion Criteria:

1. The subjects who have received radiation therapy within 4 weeks prior to randomization;
2. Those who have received hematopoietic stem cell transplantation or bone marrow transplantation
3. Patients who have been treated with G-CSF analogs or PEG-G-CSF analogs within 4 weeks prior to randomization;
4. Subjects with a history of chronic granulocytic leukemia or myelodysplastic syndromes;
5. People at high risk for ARDS;
6. Patients with unexplained splenomegaly on physical examination and/or CT scan or ultrasound, as well as any condition that may cause splenomegaly (e.g., thalassemia, glandular fever, malaria, etc.);
7. Patients who currently have or have had sickle cell anemia;
8. Those with a combined history of malignant tumors (except for the following: cured non-melanoma skin cancer, cervical cancer in situ, limited prostate cancer, superficial bladder cancer, and other malignant tumors with a disease-free survival period of more than 5 years);
9. Those diagnosed with advanced breast cancer combined with distant metastases;
10. Patients with known cerebrovascular malformations (e.g., cerebral hemangiomas), epilepsy;
11. Patients with severe mental or neurological disorders;
12. Patients with severe cardiovascular disease: history of myocardial infarction within 1 year prior to first administration of study drug; sick sinus syndrome, atrioventricular block II or greater, ventricular fibrillation, torsional ventricular tachycardia, sustained ventricular tachycardia; electrocardiogram indicative of abnormal clinically significant QRS wave lowering; congenital prolonged history of the QT interval; left ventricular ejection fraction <50%; NYHA cardiac function class III or IV; poorly controlled hypertension. Poorly controlled hypertension: blood pressure >160 mmHg systolic and/or >100 mmHg diastolic despite antihypertensive medications; congestive heart failure; stable coronary artery disease; unstable angina pectoris;
13. Liver function indexes: ALT, AST, TBIL ≥1.5 times the upper limit of normal before enrollment; Kidney function indexes: Scr ≥1.5 times the upper limit of normal;
14. Positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and peripheral blood Hepatitis B Virus (HBV) DNA test is greater than the normal range; Positive for Hepatitis C Virus (HCV); Positive for Human Immunodeficiency Virus (HIV);
15. Those with a current active infection (and a temperature ≥38°C) or who have received systemic anti-infective therapy within 72 hours prior to chemotherapy;
16. Patients with severe mouth ulcers;
17. Participated in 3 or more clinical trials of a drug within the last year, or participated in any clinical trial of a drug within the last 3 months, as a subject and actually used the test drug;
18. Hypersensitivity to the adjuvant or neoadjuvant chemotherapeutic agents used (e.g., docetaxel, epirubicin, carboplatin, cyclophosphamide) and to PEG-G-CSF and G-CSF analogs;
19. Lithium-treated patients were required during the clinical trial;
20. Alcohol-dependent individuals or those with a history of substance abuse;
21. Lactating and pregnant females and those planning a pregnancy within 6 months of the last injection of the test drug in this study;
22. Combined primary diseases of the cerebrovascular, hepatic, renal, endocrine, and hematologic systems of a severity judged by the investigator to be inappropriate for participation in this clinical trial;
23. Other patients who, in the judgment of the investigator, are not suitable subjects for this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of 4th degree neutropenia during chemotherapy cycle 1 | At the end of Cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Lowest neutrophil count during chemotherapy cycle 1; | At the end of Cycle 1 (each cycle is 21 days)
Time required for neutrophil count to recover from nadir to above 2.0 × 109/L during chemotherapy cycle 1; | At the end of Cycle 1 (each cycle is 21 days)
Duration of 4th degree neutropenia during cycles 2, 3, and 4 of chemotherapy; | At the end of cycles 2, 3, and 4 (each cycle is 21 days)
Incidence of 3rd or 4th degree neutropenia during cycles 1, 2, 3, and 4 of chemotherapy; | At the end of cycles 1, 2, 3, and 4 (each cycle is 21 days)
Duration of febrile neutropenia (FN) in cycles 1, 2, 3, and 4 of chemotherapy; | At the end of cycles 1, 2, 3, and 4 (each cycle is 21 days)
Incidence of neutropenic fever (FN) during cycles 1, 2, 3, and 4 of chemotherapy; | At the end of cycles 1, 2, 3, and 4 (each cycle is 21 days)
Incidence of infection during cycles 1, 2, 3, and 4 of chemotherapy; | At the end of cycles 1, 2, 3, and 4 (each cycle is 21 days)
Proportion of participants using antibiotics during cycles 1, 2, 3, and 4 of chemotherapy. | At the end of cycles 1, 2, 3, and 4 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China